CLINICAL TRIAL: NCT02362555
Title: The Effect of Nuchal Ligament Calcification on Cervical Function in Patients With Neck Pain
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Other Study IDs: CCH-140305
Record Dates: First submitted 2015-01-21; First posted 2015-02-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Neck Pain
Keywords: Ossification of nuchal ligament
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ossification of nuchal ligament: check neck function, radiography characteristics and complete functional disability questionnaire
  Interventions: Other: no intervention was used in this observational study
- Non ossification of nuchal ligament: check neck function, radiography characteristics and complete functional disability questionnaire
  Interventions: Other: no intervention was used in this observational study

INTERVENTIONS:
Other: no intervention was used in this observational study

SUMMARY:
Ossification of nuchal ligament often observed in patient with chronic neck pain, previous study showed ossification of nuchal ligament was associated with cervical spondylosis and radiculopathy. Patient with chronic neck pain was divided into two groups according to the presence of ossification of nuchal ligament on cervical radiographic images.

This study is to evaluate and compare the neck function including range of motion, neck strength and pressure pain threshold, radiography characteristics and functional disability between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neck pain and stiffness last for more than 1 month

Exclusion Criteria:

* cervical trauma or fracture in 3 months
* evidence of cervical spine instability
* rheumatoid cervical spondylopathy
* previous cervical surgery
* head and neck cancer
* previous radiotherapy over neck and surrounding
* those complicated with myelopathy
* contraindication to radiography like pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with chronic neck pain
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Degrees of cervical range of motion | 1 day ( first visit)
  active range of motion in flexion, extension,lateral bending and rotation direction with Cervical Range of Motion (CROM) instrument
Angles of cervical lordotic curve at C2-C7 on cervical x-ray | within one week after first visit
  measured by both modified Cobb method and Harrison posterior tangent method at C2-C7 in every participants
Scores of functional disability as a measure of effects of neck pain on daily living | 1 day ( first visit)
  neck disability index (NDI) with 10-item scaled questionnaire
The values of neck flexor, extensor, lateral bending and rotation strength | 1 day ( first visit)
  measured with a handheld dynamometer
The values of pressure pain threshold as a measure of participants' pain sensitivity | 1 day ( first visit)
  Pressure gauge algometer was applied to bilateral upper trapezius

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital Taiwan, Changhua, Taiwan